CLINICAL TRIAL: NCT03028922
Title: A Prospective, Multi-centre Study Evaluating Creos™ Xenogain Bone Graft Substitute in Horizontal Ridge Augmentation in the Premolar and Molar Region of the Mandible
Brief Title: A 1-year Clinical Investigation on the the CREOS™ XENOGAIN Bone Graft SUBSTITUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-189
Record Dates: First submitted 2017-01-10; First posted 2017-01-23 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Horizontal Bone Augmentation
Keywords: creos xenogain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- creos xenogain (Other): Patients in need of bone augmentation prior to implant insertion will undergo GBR procedure using Creos xenogain bone graft substitute
  Interventions: Device: creos xenogain

INTERVENTIONS:
Device: creos xenogain — GBR procedure will be performed using creors xenogain bone graft substitute in patients that need horizontal bone augmentation prior to implant placement. The defect should be located in the pre-molar and molar region of the mandible

SUMMARY:
This clinical investigation is a prospective, multi-centre study to evaluate bone gain after horizontal augmentation using creos xenogain bone graft substitute. Patients included in the study are in need of a GBR procedure prior to implant placement in the premolar and posterior region of the mandible.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, multi-centre study to evaluate bone gain after horizontal augmentation using creos xenogain bone graft substitute.

Patients included in the study are in need of a GBR procedure prior to implant placement in the premolar and posterior region of the mandible.

Primary endpoint include the bone gain after 8 months healing period, while secondary endpoints includes histological analysis 8 months after performance of the augmentation procedure as well as Implant survival, implant success and marginal bone levels evaluated over a period of 1 year after definitive prosthetic delivery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 80 years old.
* Patient has signed informed consent to participate in the study.
* Patients in need of horizontal ridge augmentation prior to implant placement in the premolar and posterior region of the mandible
* Horizontal defect classified as: Horizontal medium defect (Hm) (4-6 mm defect) or Horizontal large defect (Hl) (≥7 mm defect)
* Patients presented with a combination defect Horizontal/Vertical with a maximum of 2mm loss of vertical dimensions (minimal vertical dimension for patient inclusion is 7.5 mm defined as the distance from the anatomical landmark, alveolar nerve or lingual dehiscence)
* The subject must be in good physical and mental condition
* The subject is willing and able to comply with all study related procedures (such as exercising oral hygiene and attending all follow-up procedures).
* Full-mouth bleeding score (FMBS) lower than 25%.
* Full-mouth plaque score (FMPI) lower than 25%.
* The subject is suitable for a 2-stage surgical procedure

Exclusion Criteria:

* Severe bone defect classified as: Vertical medium (Vm) (4-6 mm defect) or Vertical large, (Vl) (≥7 mm)
* Medium (Cm) and Large (Cl) classified combination defects Prior bone augmentation in the area planned for treatment (i.e ridge preservation)
* Health conditions, which do not permit the surgical (including anesthesia) or restorative procedure.
* Any disorders directly in the planned implant area such as previous tumors, chronic bone disease.
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc).
* Alcohol or drug abuse as noted in subject records or in subject history.
* Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or history.
* Heavy smoking (> 10 cigarettes per day).
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake or A1c level above 8%.
* Poor compliance.
* Active periodontal disease involving the residual dentition.
* Mucosal diseases in the areas to be treated.
* Pregnant or lactating women at the time of bone augmentation procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-04 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Bone gain 8 months after bone augmentation procedure for implant placement. | 8 months
  To evaluate bone gain 8 months after bone augmentation procedure for implant placement.

SECONDARY OUTCOMES:
Implant survival | 6 months and 1 year after definitive prosthetic delivery
  To demonstrate cumulative survival rate of the implants placed in the augmented bone at 6 months and at 1 year after definitive prosthetic delivery.
Implant success | 6 months and 1 year after definitive prosthetic delivery
  To demonstrate cumulative success rate of the implants placed in the augmented bone at 6 months and 1 year after definitive prosthetic delivery.
Marginal bone levels | 6 months and 1 year after definitive prosthetic delivery
  To demonstrate the changes in marginal bone levels (ΔMBL) around the implants placed in the augmented bone as measured and evaluated by periapical films, 6 months and 1 year after definitive prosthetic delivery
Histological analysis prior to implant insertion including percentage of vital bone, residual graft and connective tissue or other non bone components | 8 months
  A bone sample using a trephine bur will be collected after 8 months and prior to implant insertion in order to perform histological analysis. The analysis will include the following parameters: percentage of vital bone and residual graft and connective tissue and if present other non bone components
Soft tissue outcome 1 year after definitive prosthetic delivery | 1 year
  Soft tissue outcome is a combination of different parameters that include gingival index, bleeding index, keratinized mucosa and pink esthetic score
oral health related quality of life assessment | 1 year
  To demonstrate pre- and postoperatively the oral health related quality of life assessment using the Oral Health Impact Profile questionnaire (OHIP-14).

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (2):
  - Praxisklinik der Zahnheilkunde am Luisenhospital, Aachen
  - Universitäts Klinikum Frankfurt, Frankfurt
- Italy (2):
  - Clinica Odontoiatrica - Dipartimento di Neuroscienze, Università di Padova, Padua
  - Clinica Merli, Rimini
- Serbia (2):
  - Military Academy of Belgrade, Oral Surgery, Belgrade
  - University of Belgrade, Periodontology, Belgrade

REFERENCES:
- [Derived] Lorenz J, Ghanaati S, Aleksic Z, Milinkovic I, Lazic Z, Magic M, Wessing B, Grotenclos RS, Merli M, Mariotti G, Bressan E, De Stavola L, Sader R. Horizontal Guided Bone Regeneration of the Posterior Mandible to Allow Implant Placement: 1-Year Prospective Study Results. Clin Oral Implants Res. 2025 Jan;36(1):100-116. doi: 10.1111/clr.14363. Epub 2024 Oct 1. PMID 39351703